CLINICAL TRIAL: NCT04411719
Title: Prognosis of Acute DOC
Brief Title: Outcome Prediction in Patients With Acute Disorders of Consciousness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Outcome in DOC
Record Dates: First submitted 2020-05-28; First posted 2020-06-02 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-05

CONDITIONS: Consciousness Disorder
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EEG and Microexpression Analysis: Participants will be acutely unresponsive ICU patients. They will undergo non-invasive observational procedures, including EEG monitoring during exposure to emotional auditory stimuli, and concurrent video recording for microexpression analysis. Patient outcomes will be assessed at three, six, and twelve-month intervals post-initial observation.

SUMMARY:
Prior research has indicated a link between outcomes in patients with disorders of consciousness (DOC) and their responses to emotional auditory stimuli. Given the high degree of uncertainty in acute situations, this study plans to record EEG responses and observe microexpressions in DOC patients during exposure to auditory stimuli, with the aim to identify more reliable prognostic indicators. The goal is to uncover potential patterns or signals that can contribute to a more comprehensive understanding of a patient's condition, and thereby provide more accurate prognostication.

DETAILED DESCRIPTION:
This study intends to probe the potential of electroencephalography (EEG) and microexpression analysis for predicting the outcomes of acutely unresponsive patients within the intensive care unit (ICU). Previous research has illuminated a relationship between patients' emotional responses to auditory stimuli and their prognosis. However, the predictive utility of these responses in the context of acute conditions remains largely unexplored.

At the onset of the study, participants will undergo EEG monitoring while exposed to a pre-determined set of emotional auditory stimuli. Additionally, the patients' facial expressions will be captured via video for subsequent microexpression analysis.

Follow-up assessments of the patients' status will be conducted at three, six, and twelve-month intervals. Using cutting-edge analytical techniques, the goal is to decode these EEG and microexpression responses. This study aims to identify possible correlations between these findings, the patients' diagnoses, and their respective outcomes over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute brain injury (<28 days) in ICU
* GCS ≤ 8
* ≥ 2 days after sedation
* Normal hearing, with auditory startle reflex

Exclusion Criteria:

• Children under 18

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Unresponsive patients after severe brain injury.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale-Extended (GOS-E) | Month 1
  GOS-E is an extended version of the Glasgow Outcome Scale (GOS), which was developed to provide a more detailed assessment of patient functionality and quality of life after experiencing such an injury. It has eight categories: Dead, Vegetative State, Lower Severe Disability, Upper Severe Disability, Lower Moderate Disability, Upper Moderate Disability, Lower Good Recovery, and Upper Good Recovery.
Glasgow Outcome Scale-Extended (GOS-E) | Month 3
  GOSE will be assessed 3 months after brain injury.
Glasgow Outcome Scale-Extended (GOS-E) | Month 6
  GOSE will be assessed 6 months after brain injury.
Glasgow Outcome Scale-Extended (GOS-E) | Month 12
  GOSE will be assessed 12 months after brain injury.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Prof, Dr, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No